CLINICAL TRIAL: NCT03643913
Title: The Effect of Deep Neuromuscular Block and Reversal With Sugammadex on Surgical Conditions and Perioperative Morbidity in Shoulder Surgery Using a Deltopectoral Approach
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: MSD Belgium BVBA (Industry)
Responsible Party: Principal Investigator, Harm Hoekstra, prof. dr., Prof. Dr. Harm Hoekstra, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NS918
Record Dates: First submitted 2018-08-06; First posted 2018-08-23 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Shoulder Pain; Anesthesia
MeSH Terms: conditions — Shoulder Pain | interventions — Neuromuscular Blocking Agents

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The patient and the surgeon are blinded for the intervention. The anesthesist knows the allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Comparison group (Active Comparator): Neuromuscular Blocking Agents and reversing agents: The comparison group will receive anesthesia top up Esmeron dose to maintain a Train Of Four (TOF) count of maximum 2 during the whole procedure. This represents moderate neuromuscular block conditions. A neuromuscular monitor (PHILIPS integrated) will be used to evaluate TOF count.
  To maintain TOF at 2 and according to our practice a bolus injection of 0,1 mg/kg Rocuronium will be given when TOF count returns to 3. This dose will be repeated if TOF does not go back to 2 within 2 minutes after bolus injection. TOF guard and TOF tube will be used at the ulnar nerve at the contralateral side and will be checked continuously during surgery.
  Reversal of the TOF=2 will be done by Sugammadex 2 mg/kg at end of procedure (Time of last suture)
  Interventions: Procedure: Moderate neuromuscular block; Drug: Neuromuscular Blocking Agents and reversing agents
- Deep group (Experimental): Neuromuscular Blocking Agents and reversing agents: The deep group will receive deep neuromuscular block, using a infusion of Esmeron at 0,1mg/kg/hour. A post tetanic count will be performed and our target will be to have a PTC 1-2. The standard infusion will be adjusted as such. Reversal will be achieved by Sugammadex 4 mg/kg depending on reversal speed at the end of procedure (Time of last suture)
  Interventions: Procedure: Deep neuromuscular block; Drug: Neuromuscular Blocking Agents and reversing agents

INTERVENTIONS:
Procedure: Deep neuromuscular block — Deep neuromuscular block requiring higher doses of Esmeron to target a post tetanic count (PTC) of 1-2 and higher doses of Bridion to reverse the block (4mg/kg).
  Arms: Deep group
Procedure: Moderate neuromuscular block — Normal neuromuscular block requiring dosis of Esmeron to target a train of four (TOF) count of max 2 and lower doses of Bridion to reverse the block (2mg/kg).
  Arms: Comparison group
Drug: Neuromuscular Blocking Agents and reversing agents — Deep neuromuscular block versus moderate neuromuscular block.

SUMMARY:
The study evaluates wether deep neuromuscular block during entire surgical procedure to the gleno-humeral joint or the proximal humerus using a deltoideo-pectoral approach results in less muscular damage to the deltoid muscle and therefore less post-operative pain and an earlier functional recovery..

ELIGIBILITY:
Inclusion Criteria:

• Adult patient undergoing elective or semi-elective surgery to the gleno-humeral joint or the proximal humerus using a deltoideo-pectoral approach

Exclusion Criteria:

* Inability to consent because of mental status
* Open injuries involving the deltoid muscle
* Previous open surgery on the shoulder joint.
* American Society of Anaesthesiologists (ASA) physical status >II
* Age <18 or >85 year old
* Body mass index (BMI) <18.5 or >35 kg/m2
* Renal insufficiency (glomerular filtration rate <40 ml/min)
* Impaired liver function (hepatic cirrhosis, cholestatic jaundice)
* Neuromuscular disease
* Pregnancy
* Breastfeeding
* Predicted difficult airway
* Patients receiving medications known to interact with neuromuscular blocking agents
* Allergy to any drug included in the anesthetic protocol

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2024-11-27 (Actual)

PRIMARY OUTCOMES:
Modified Leiden score | 1 Day of surgery
  the surgeon will be asked to score the surgical conditions on a five step scale based upon previously used scales:
  * grade 5: optimal surgical conditions, perfect access to the proximal humerus, glenohumeral joint and excellent visibility.
  * grade 4: good conditions: adequate surgical conditions to perform the surgery, but not optimal
  * grade 3: acceptable conditions, surgical procedure is jeopardized, but adequate surgical result is obtained, eventually after additional intervention
  * grade 2: poor conditions, exposure and handling hindered resulting in suboptimal surgical outcome
  * grade 1: extremely poor conditions, the surgeon is unable to work because of the inability to get access to the shoulder joint because of inadequate muscle relaxation.
Visual analogue scale (VAS) | Day 3 post-operative at 14 o' clock
  Scale ranges from 0 to 10 representing respectively no pain and wordt imaginable pain.

SECONDARY OUTCOMES:
Muscular damage | 1 Day of surgery
  Two light photos will be taken before closure of the deltoideopectoral interval to document the muscular damage by the surgeon using a grading score (1-4, 1=no muscular damage, 2=superficial damage (fraying) or contusion, 3=muscular tear < 1 cm depth, 4=muscular tear > 1 cm depth).
Muscular damage | 1 year after inclusion
  Two light photos will be taken before closure of the deltoideopectoral interval to document the muscular damage by two independent reviewers (surgeons blinded to the procedure) using a grading score (1-4, 1=no muscular damage, 2=superficial damage (fraying) or contusion, 3=muscular tear < 1 cm depth, 4=muscular tear > 1 cm depth).
VAS | The scoring will be done at 8-14 and 20 o'clock on days 1-3-5 post-operative and once a day from day 5 to day 30 post-operative.
  Scale ranges from 0 to 10 representing respectively no pain and worst imaginable pain. Post-operative pain will be scored using a VAS-pain scale ranging from 0 (no pain) to 10 (worst imaginable pain).
Analgesic needs | Up to 5 days post-operative
  The analgesic needs of the patient during hospitalization will be derived from the Electronic Medical Prescription (EMV) module of the Electronic patient file system. The total morphine consumption will be assessed in all groups as well as rescue medication such as ketalar, NSAID's catapressan and paracetamol.
Analgesic needs | From hospital discharge to 30 days post-operative
  The analgesic needs of the patient after hospitalization will be derived from a patient diary.
Length of stay at post-anesthesia care unit (PACU) | 1 Day of surgery
  Evaluation and length of stay at the PACU will also be examined as this clearly reflects the amount of post-operative comfort or possible adverse effects witnessed post procedure. The parameter will be expressed in hours and there will be two measurement. The time of expected discharge and the actual discharge (with reasons of possible delay between those two figures expressed in minutes or hours).
Length of surgery | intraoperative
  Will be expressed in %. As different procedures are being performed within this study, absolute length would not be indicative for ease of procedure. Therefore we express length of surgery as actual length of the procedure (incision to closure), divided by the mean length of the 10 last identical procedures (out of the study) performed by the same surgeon.
Length of stay | from day 3 up to 3 weeks after surgery
  Is defined as post-operative length of stay, the day of surgery being day 0. This parameter will be expressed in days. As post-operative pain is one of the principal reasons for hospitalization after shoulder surgery, we believe this parameter is an indirect measure for post-operative pain.
Evaluation of dry catheter technique | 1 Day of surgery
  Evaluation of the efficacy of the catheter will be done 30 minutes after the bolus injection. Efficacy will be tested by using ether swab to test sensory block and also motorfunction evaluation of the motorjoint (raising arm to full height pass/fail).

CONTACTS AND LOCATIONS:
Overall Officials: Harm Hoekstra, Prof. Dr., Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No